CLINICAL TRIAL: NCT06639789
Title: Evaluation of the Effect of a New Formulation of Vitamin B12 on Physical and Mental Performance in Trained Cyclists.
Brief Title: Effect of a New Formulation of Vitamin B12 on Physical and Mental
Acronym: PERB12
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Javier Martínez Noguera (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, PhD (Head of the nutrition area of the Research Center for High Performance Sport), Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CE052416
Record Dates: First submitted 2024-09-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Performance Enhancing Product Use
Keywords: Anaerobic performance; Power; Mental fatigue; Vitamins; Recovery
MeSH Terms: conditions — Mental Fatigue | interventions — Vitamin B 12

STUDY DESIGN:
Intervention Model Description: A randomized crossover study will be conducted in which 18 subjects will perform the following conditions: B12) 1 mg/d vitamin B12; PLA) 200 mg/d placebo (microcrystalline cellulose) 3 days before physical and cognitive performance tests.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B12 (B12) (Experimental): Subjects in this group will intake 1 mg/day of vitamin B12 three days before the tests.
  Interventions: Dietary Supplement: Vitamin B12 (B12)
- PLACEBO (PLA) (Placebo Comparator): Subjects in this group will intake 200 mg/day of microcrystalline cellulose three days before the tests.
  Interventions: Dietary Supplement: PLACEBO (PLA)

INTERVENTIONS:
Dietary Supplement: Vitamin B12 (B12) — The new formulation of vitamin B12 will be ingested 3 days before and on the day of testing (3 hours before).
  Arms: Vitamin B12 (B12)
Dietary Supplement: PLACEBO (PLA) — The placebo will be ingested 3 days before and the same day of the tests (3 hours before).
  Arms: PLACEBO (PLA)

SUMMARY:
This clinical study evaluates the effect of acute intake of a new vitamin B12 formulation on anaerobic and cognitive performance variables. One of the limiting factors for the potential beneficial effects of vitamin B12 is its bioavailability. This new formula improves this aspect, so that by improving plasma levels of B12 we will be able to relate whether this situation may be related to improved performance or cognitive tasks.

DETAILED DESCRIPTION:
Participants

All participants were informed about the procedures and provided signed informed consent. The study was conducted in accordance with the guidelines of the Declaration of Helsinki Declaration for Research Involving Human Subjects and the protocol was approved by the Institutional Review/Ethics Committee of the Catholic University of Murcia (Code: CE052416).

Study design

Randomized, double-blind, placebo-controlled, crossover clinical trial with 2 study groups (vitamin B12 and placebo). Cyclists were instructed to take the supplement (vitamin B12 or placebo) with breakfast on the three days before the tests and 3h before the test day, and to continue with their usual diet and training programme. Subjects in both groups were instructed not to consume vitamin B12-rich foods for 7 days before and during the study. Between each intervention (B12 and Placebo) there was a 7-day washout period.

Procedures

Participants visited the laboratory on three occasions. Visit 1 consisted of a medical examination and a blood draw to determine health status. At visits 2 and 3, a 24-hour diet reminder and a Wingate test, mental fatigue test and venous blood draw were performed. The sports nutritionist prescribed a standardized breakfast before each testing session (visits 2 and 3).

Pre- and post-evaluation test

Visit 1:

Health status blood test: A general blood test will be performed both pre- and post-supplementation. The blood will be drawn through a vein (fasting).

Medical examination: A medical history of family and personal history, an electrocardiogram (ECG) at rest and a medical examination (auscultation, blood pressure, etc.) will be carried out to certify that the person is healthy and does not present a risk to participate in the study (Fasting).

Body composition by absorptiometric densitometry (DXA): A body composition test will be performed using the double energy absorptiometric densitometry technique (X-rays), with the aim of determining parameters of fat mass, fat-free mass and fat percentage. In addition, anthropometry will also be used to determine changes in body composition (fat and muscle mass) (Fasting).

Visits 2 and 3:

Anaerobic power and mechanical power output: After a standardised breakfast, a Wingate test was performed on a cycle ergometer. The Wingate test (WAnT) consisted of a 30 s sprint on a cycle ergometer (Monark Ergomedic 894E Peak Bike, Vansbro, Sweden). Breaking strength was held constant at 7.5% of each individual's body mass. All participants were verbally encouraged to pedal as fast as possible throughout the sprint.

Mental fatigue test: All participants will be tested for the evaluation of reaction time to a sequence of lights set by the investigator before and after the performance test.

Biochemical markers: A venous blood draw will be performed by medical personnel before and after the performance test, in which vitamin B12, creatine kinase and lactate dehydrogenase levels will be analyzed.

All data of the subjects who participated in the study were stored in a computer system with a security key. In addition, some of the data was also recorded on paper and kept under lock and key, accessible only to the researchers of this project.

ELIGIBILITY:
Inclusion Criteria:

* Male cyclists who have competed in both junior and amateur categories.
* Cycling between 6-15 hours of training per week.
* BMI between 18-25 kg/m2.

Exclusion Criteria:

* Smokers or regular alcohol drinkers.
* Persons suffering from a metabolic, cardiorespiratory or digestive pathology or anomaly.

digestive system.

* People who have suffered an injury in the last 6 months that limits the performance of the study tests. of the study tests.
* People taking supplements or medication in the 2 weeks before the start of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wingate test | Throughout study completion, an average of 3 weeks
  This test consists of 5 efforts of 30 seconds at maximum intensity with a recovery of 3 minutes on a bike. In this test the peak and average power of each effort and the total average will be evaluated. In addition, the time to maximum peak power and the fatigue index.

SECONDARY OUTCOMES:
Mental fatigue test | Throughout study completion, an average of 3 weeks
  In this test, we will measure the speed of reaction in the resolution of a sequence of lights set by the researcher before and after the end of the performance test.
Biochemical markers | Throughout study completion, an average of 3 weeks
  Vitamin B12, creatine kinase and lactate dehydrogenase concentrations are also measured before and after the performance tests.
Sleep Quality Questionnaire (Pittsburgh) | Throughout study completion, an average of 3 weeks
  The questionnaire will be carried out 3 days before and one day after the performance tests.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier J Martínez Noguera, Study Chair — Research Center for High Performance Sport. Catholic University of Murcia
Locations (1):
- Research Center for High Performance Sport. Catholic University of Murcia, La Ñora, Murcia, Spain